CLINICAL TRIAL: NCT01454479
Title: A Phase I Study of Lapatinib (Tykerb) Plus Ixabepilone (Ixempra) as 2nd-line Treatment for Patients With HER-2 Overexpressed Recurrent or Persistent Endometrial Carcinoma or Carcinosarcoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hung-Hsueh Chou (Other)
Collaborators: GlaxoSmithKline (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Hung-Hsueh Chou, Principal Investigator of Gyncological department, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-3771A3
Record Dates: First submitted 2011-09-28; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Recurrent Endometrial Cancer
Keywords: Lapatinib; Ixabepilone; HER-2; Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Lapatinib; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib (Tykerb) Plus Ixabepilone (Experimental)
  Interventions: Drug: Lapatinib and ixempra

INTERVENTIONS:
Drug: Lapatinib and ixempra — Ixabepilone 40 mg/m2 Lapatinib 250 mg
  Other Names: Lapatinib; Ixempra

SUMMARY:
Endometrial cancer (EC) is the 8th most common female cancer in Taiwan. Its incidence is increasing in the recent few years, around 1,200 new cases per year. The outcome of recurrent EC is disappointing, except focal recurrences that could be irradiated or removed. Chemotherapy is currently the most common salvage treatment for recurrent endometrial cancer. However, the response rate (RR) to 2nd-line treatment is approximately 0-27.3%, with short median time to progression, 2-3.9 months and low overall survival, 6.4-11 months.

Due to progress of studies on the molecular and genetic basis of cancer and cellular signaling pathways, targeted therapy has been developed for various cancer treatments. A Gynecologic Oncology Group study found 44% of advanced endometrial cancer had HER>=2+ and the ratio of HER2:chromosome 17 (CEP17) >=2. Another study showed that HER>=2+ was seen in 47% of carcinosarcoma. These evidences indicated HER2 gene amplification and HER2 overexpression occur in endometrial cancer and carcinosarcoma, especially in those of high grade and recurrence. Lapatinib (L), an oral inhibitor of both EGFR(epidermal growth factor receptor) and HER2(human epidermal growth receptor), has been shown to be an effective treatment in HER2/neu overexpressing metastatic breast cancer. Ixabepilone is a semisynthetic analog of the natural product epothilone B, and recently has been approved by US Food and Drug Administration as a treatment option in metastatic breast cancer. It was also observed that lapatinib + ixabepilone killed more breast tumor cells than trastuzumab + paclitaxel in vitro. Two GOG(Gynecologic Oncology Group) studies had reported that weekly Ixabepilone as 2nd-line chemotherapy provided a similar RR to 3-weekly regimen of 14.3% in platinum- and taxane-resistant epithelial ovarian cancer with less severe toxicities. The combination of lapatinib and ixabepilone is expected to become an effective treatment for recurrent endometrial cancer and carcinosarcoma, but the ideal dose is yet to be surveyed.

DETAILED DESCRIPTION:
Patients receive weekly Ixabepilone 32 mg/m2 (D1) and a 4-level of oral Lapatinib 500-1250 mg once daily continuously. The recommended duration of treatment for each patient 21 days a cycle of total 6 cycles or until disease progression, or unacceptable toxicity or patient's refusal occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed carcinoma or carcinosarcoma of the endometrium with evidence of persistent disease or progression after initial surgery and adjuvant chemotherapy, radiotherapy, or both, not amenable for curative salvage therapy.
2. ErbB2 gene amplification by FISH (ErbB2 gene copies to chromosome 17 signals) of > = 2.0; ErbB2 overexpression is defined by immunostaining >=2 for ErB2
3. Measurable disease, defined as ≥1 lesions that can be accurately measured in

   * 1 dimensions as ≥20 mm by conventional techniques OR as ≥10 mm by spiral CT scan, MRI or PET scan (those who undergo cytoreductive salvage surgery with residual tumor ≥ 20 mm are eligible)
4. Those who are chemotherapy-naive be enrolled until failing one chemotherapy regimen
5. Prior treatments with radiation therapy for palliative management of metastatic disease is permitted provided that at least 4 weeks have elapsed since the last fraction of radiation therapy, disease progression has been documented and all treatment related adverse events are ≦ grade 2 at the time of registration.
6. Life expectancy ≥ 12 weeks
7. ECOG(Eastern Cooperative Oncology Group) performance status 0-2
8. Patients must have normal organ and marrow function measured within 14 days

Exclusion Criteria:

1. Previously unirradiated, isolated vaginal, pelvic or paraaortic lymph node, lung (which confined to one lobe that can be resected or radiated) recurrence or other potentially curable recurrence such as central pelvic recurrence for which a pelvic exenteration is feasible
2. Pregnant or lactating women.
3. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
4. Prior therapy with Lapatinib or Ixabepilone.
5. CNS metastases.
6. Ongoing other concurrent investigational agents or anticancer therapy
7. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious non- healing wound/ulcer/bone fracture, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
9. Preexisting peripheral neuropathy≥G2

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dosage (MTD) of the combination of lapatinib with Ixabepilone as 2nd-line chemotherapy in patients with treatment in HER2 overexpressed recurrent or persistent endometrial cancer or carcinosarcoma | 2013/Apr
  Determine the Maximum Tolerated Dosage (MTD) of the combination of lapatinib with Ixabepilone as 2nd-line chemotherapy in patients with treatment in HER2 overexpressed recurrent or persistent endometrial cancer or carcinosarcoma.